CLINICAL TRIAL: NCT02377388
Title: DPP-4 Inhibitors in Patients With Type 2 Diabetes and Acute Myocardial Infarction:Effects on Platelet Function
Brief Title: DPP-4 Inhibitors and Acute Myocardial Infarction:Effects on Platelet Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of São Paulo GH
Record Dates: First submitted 2015-01-05; First posted 2015-03-03 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-02

CONDITIONS: Platelet Aggregation During Acute Myocardial Infarction
Keywords: diabetes mellitus; platelet function testing; acute coronary syndromes; saxagliptin; sitagliptin; dpp-4 inhibitors
MeSH Terms: conditions — Diabetes Mellitus; Acute Coronary Syndrome | interventions — Sitagliptin Phosphate; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment: DPP4 -i (Active Comparator): Use of DPP4-i :
  sitagliptin 50 mg (if glomerular filtration rate-GFR <50 ml/min at randomization) or 100 mg (if GFR>50 ml/min at randomization),during 30 days,once-daily(OD)
  OR
  saxagliptin 2,5 mg (if glomerular filtration rate-GFR <50 ml/min at randomization) or 5 mg (if GFR>50 ml/min at randomization),during 30 days,once-daily(OD)
  Interventions: Drug: sitagliptin OR saxagliptin
- control (Placebo Comparator): placebo tablets identical to active comparator,administered according to GFR at randomization,during 30 days,OD
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sitagliptin OR saxagliptin — sitagliptin OR saxagliptin tablets, 48(+-24) hours after the beginning of an AMI,and both arms in use of dual anti-platelet therapy (DAPT) .
  Other Names: januvia ® OR onglyza ®
  Arms: treatment: DPP4 -i
Drug: placebo — placebo tablets, 48(+-24) hours after the beginning of an AMI,and both arms in use of dual anti-platelet therapy (DAPT) .
  Other Names: PBO
  Arms: control

SUMMARY:
Cardiovascular events are the main cause of mortality in diabetic patients ,on the other hand,during an acute myocardial infarction(AMI),hyperglycemia increases mortality and is related to different pathophysiologic processes.

More important evidence regarding the effect of glycemic control on AMI patients prognosis is contradictory,and the potential benefits of dipeptidyl peptidase-4 inhibitors(DPP4-i) in this setting is unknown.

The aim of this study is to assess the presence of pleiotropic effects of DPP4-i(sitagliptin or saxagliptin) and their relationship with glycemic control during in-hospital phase of AMI.

DETAILED DESCRIPTION:
Randomized clinical trial,double-blinded,placebo-controlled, in a single center, to assess the influence of DPP4-i on platelet aggregability in type 2 diabetic patients with acute myocardial infarction in use of dual anti platelet therapy (DAPT) .

Others exploratory analysis include:glycemic control ,infarct size,genetic analysis and cholesterol metabolism.

After giving signed informed consent,eligible subjects will be randomly allocated to receive saxagliptin or placebo, in the first 48 hours (+-24) after the beginning of an AMI.

The investigator and subjects will be blinded to trial treatment,and a person not involved in trial conduct will prepare the doses of study drug.The doses will be administered by mouth,in a once daily basis by the investigator.

Blood samples will be collected by the investigator according to pre-specified outcomes and time frames.

Evaluation of glycemic control by CGM will be carried out by the investigator,including insert and withdrawal of the device.

Treatment of the acute event,(AMI) will be done according to routine procedures from coronary care unit.

Serious adverse event report taking into consideration all-cause mortality, cardiovascular mortality, hospitalization for heart failure and pancreatitis, will be done according to presence of these events.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of type 2 diabetes mellitus,with treatment including insulin and/or oral antidiabetic agent;
* subjects without previous diagnosis of diabetes,but HbA1c admission >= 6,5% during current hospital-stay
* AMI with or without ST-elevation;
* use of double antiplatelet therapy;
* signed informed consent term

Exclusion Criteria:

* GFR <30 ml/min;
* use of DPP4 inhibitors or glucagon- like peptide-1(GLP1) analogue in the past 6 months;
* use of strong inhibitors of cytochrome P450(CYP3A4/5) ou glucocorticoids;
* severe systemic decompensation requiring insulin infusion;
* Killip classification of myocardial infarction grade >2;
* previous history of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
changes on platelet aggregability. | baseline and 4(+-2) days after drug exposure.
  Comparison on platelet function between two therapeutic arms in a double-blind randomized fashion. Platelet aggregability will be measured 4(+-2) days after drug exposure,using a point-of-care test (VerifyNow Aspirin) in type 2 diabetic patients with AMI on dual antiplatelet therapy (ASA+ ticagrelor or clopidogrel according to institutional routine).

SECONDARY OUTCOMES:
changes on platelet aggregability. | baseline and 30(+-5) days after drug exposure.
  Primary outcome measure analyzed at baseline and 30(+-5) days after drug exposure.
platelet aggregability differences by two point-of-care methods. | baseline and 4 (+-2) days after drug exposure.
  Comparison on platelet aggregability by two different methods :Verify Now and Multiplate.
platelet aggregability differences by two point-of-care methods. | baseline and 30(+-5) days after drug exposure.
  Comparison on platelet aggregability by two different methods (Verify Now and Multiplate .

OTHER OUTCOMES:
changes in glycemic control(glycemic variability assessed by standard deviation(SD) of capillary glucose samples). | baseline up to 1 week.
  Evaluated by measurements of capillary glucose samples by point-of care test during the length of coronary care unit(CCU) stay( expected average of 1 week).The glycemic variability will be obtained by calculating the standard deviation(SD).
changes in glycemic control(glycemic variability assessed by continuous glucose monitoring system - CGM). | baseline and 48 (+-24) hours after drug exposure.
  Evaluated by mean amplitude of glycemic excursions(MAGE) by the use of CGM
changes on platelet aggregability on pre-specified subgroups. | baseline and 4 (+-2)days after drug exposure.
  Changes on platelet aggregability will be compared on pre-specified subgroups:
  elderly (age >65 yrs-old) versus non-elderly;
  male versus female;
  smoking versus non-smoking patients;
  obese(BMI>30 Kg/m2) versus non-obese;
  length of diabetes;
  baseline glucose;
  glycated hemoglobin(HbA1c) < 9% and >9 %
rate of hypoglycemia during coronary care unit stay. | baseline up to 1 week .
  Rate of capillary glucose <70 mg/dL and <40 mg/dL,evaluated by capillary glucose measurements by point-of-care tests,during CCU stay(expected average of 1 week).
total of insulin doses requirement during coronary care unit stay. | baseline up to 1 week .
  Comparison of the total requirement of correctional insulin between treatment and control arms after drug exposure.
incidence of composite end-point. | baseline and 30 (+-5) days after drug exposure
  Comparison the incidence of composite end-point between two arms.Composite end-point include:
  cardiovascular death;
  unstable angina;
  stroke ;
  hospitalization for heart failure;
  new non fatal myocardial infarction ;
  coronary revascularization .
Infarct size. | baseline up to 1 week
  Analysis of infarct size between two arms, by peak of creatine kinase(CK-MB) during CCU stay(expected average of 1 week).
cholesterylester transfer protein(CETP) mass | baseline
  Analysis of CETP mass between two arms.
measure of safety, Number of participants with adverse effects by analysis on changes of serum level | baseline and 30(+-5) days after drug exposure.
  Number of participants with adverse effects by analysis on changes of serum level of :
  alanine transferase;
  brain natriuretic peptide(BNP);
  amylase;
  lipase.

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Nicolau, MD,PhD, Principal Investigator — Heart Institute(InCor)-University of São Paulo GH-Medical School
Locations (1):
- Heart Institute(InCor)-Acute Coronary Care Unit, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kosiborod M, Rathore SS, Inzucchi SE, Masoudi FA, Wang Y, Havranek EP, Krumholz HM. Admission glucose and mortality in elderly patients hospitalized with acute myocardial infarction: implications for patients with and without recognized diabetes. Circulation. 2005 Jun 14;111(23):3078-86. doi: 10.1161/CIRCULATIONAHA.104.517839. Epub 2005 Jun 6. PMID 15939812
- [Background] Kosiborod M, Inzucchi SE, Krumholz HM, Xiao L, Jones PG, Fiske S, Masoudi FA, Marso SP, Spertus JA. Glucometrics in patients hospitalized with acute myocardial infarction: defining the optimal outcomes-based measure of risk. Circulation. 2008 Feb 26;117(8):1018-27. doi: 10.1161/CIRCULATIONAHA.107.740498. Epub 2008 Feb 11. PMID 18268145
- [Background] Goyal A, Mahaffey KW, Garg J, Nicolau JC, Hochman JS, Weaver WD, Theroux P, Oliveira GB, Todaro TG, Mojcik CF, Armstrong PW, Granger CB. Prognostic significance of the change in glucose level in the first 24 h after acute myocardial infarction: results from the CARDINAL study. Eur Heart J. 2006 Jun;27(11):1289-97. doi: 10.1093/eurheartj/ehi884. Epub 2006 Apr 12. PMID 16611669
- [Background] Nicolau JC, Maia LN, Vitola JV, Mahaffey KW, Machado MN, Ramires JA. Baseline glucose and left ventricular remodeling after acute myocardial infarction. J Diabetes Complications. 2007 Sep-Oct;21(5):294-9. doi: 10.1016/j.jdiacomp.2006.01.003. PMID 17825753
- [Background] Nicolau JC, Serrano CV Jr, Giraldez RR, Baracioli LM, Moreira HG, Lima F, Franken M, Kalil R, Ramires JA, Giugliano RP. In patients with acute myocardial infarction, the impact of hyperglycemia as a risk factor for mortality is not homogeneous across age-groups. Diabetes Care. 2012 Jan;35(1):150-2. doi: 10.2337/dc11-1170. Epub 2011 Oct 25. PMID 22028280
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Esposito K, Nappo F, Marfella R, Giugliano G, Giugliano F, Ciotola M, Quagliaro L, Ceriello A, Giugliano D. Inflammatory cytokine concentrations are acutely increased by hyperglycemia in humans: role of oxidative stress. Circulation. 2002 Oct 15;106(16):2067-72. doi: 10.1161/01.cir.0000034509.14906.ae. PMID 12379575
- [Background] Standl E, Schnell O, Ceriello A. Postprandial hyperglycemia and glycemic variability: should we care? Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S120-7. doi: 10.2337/dc11-s206. PMID 21525442
- [Background] Hermanides J, Vriesendorp TM, Bosman RJ, Zandstra DF, Hoekstra JB, Devries JH. Glucose variability is associated with intensive care unit mortality. Crit Care Med. 2010 Mar;38(3):838-42. doi: 10.1097/CCM.0b013e3181cc4be9. PMID 20035218
- [Background] Krinsley JS. Glycemic variability: a strong independent predictor of mortality in critically ill patients. Crit Care Med. 2008 Nov;36(11):3008-13. doi: 10.1097/CCM.0b013e31818b38d2. PMID 18824908
- [Background] Lipska KJ, Venkitachalam L, Gosch K, Kovatchev B, Van den Berghe G, Meyfroidt G, Jones PG, Inzucchi SE, Spertus JA, DeVries JH, Kosiborod M. Glucose variability and mortality in patients hospitalized with acute myocardial infarction. Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):550-7. doi: 10.1161/CIRCOUTCOMES.111.963298. Epub 2012 Jun 12. PMID 22693348
- [Background] Siegelaar SE, Kerr L, Jacober SJ, Devries JH. A decrease in glucose variability does not reduce cardiovascular event rates in type 2 diabetic patients after acute myocardial infarction: a reanalysis of the HEART2D study. Diabetes Care. 2011 Apr;34(4):855-7. doi: 10.2337/dc10-1684. PMID 21447661
- [Background] Malmberg K, Ryden L, Efendic S, Herlitz J, Nicol P, Waldenstrom A, Wedel H, Welin L. Randomized trial of insulin-glucose infusion followed by subcutaneous insulin treatment in diabetic patients with acute myocardial infarction (DIGAMI study): effects on mortality at 1 year. J Am Coll Cardiol. 1995 Jul;26(1):57-65. doi: 10.1016/0735-1097(95)00126-k. PMID 7797776
- [Background] Malmberg K, Ryden L, Wedel H, Birkeland K, Bootsma A, Dickstein K, Efendic S, Fisher M, Hamsten A, Herlitz J, Hildebrandt P, MacLeod K, Laakso M, Torp-Pedersen C, Waldenstrom A; DIGAMI 2 Investigators. Intense metabolic control by means of insulin in patients with diabetes mellitus and acute myocardial infarction (DIGAMI 2): effects on mortality and morbidity. Eur Heart J. 2005 Apr;26(7):650-61. doi: 10.1093/eurheartj/ehi199. Epub 2005 Feb 23. PMID 15728645
- [Background] de Mulder M, Umans VA, Cornel JH, van der Zant FM, Stam F, Oemrawsingh RM, Akkerhuis KM, Boersma E. Intensive glucose regulation in hyperglycemic acute coronary syndrome: results of the randomized BIOMarker study to identify the acute risk of a coronary syndrome-2 (BIOMArCS-2) glucose trial. JAMA Intern Med. 2013 Nov 11;173(20):1896-904. doi: 10.1001/jamainternmed.2013.10074. PMID 24018647
- [Background] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Background] Griesdale DE, de Souza RJ, van Dam RM, Heyland DK, Cook DJ, Malhotra A, Dhaliwal R, Henderson WR, Chittock DR, Finfer S, Talmor D. Intensive insulin therapy and mortality among critically ill patients: a meta-analysis including NICE-SUGAR study data. CMAJ. 2009 Apr 14;180(8):821-7. doi: 10.1503/cmaj.090206. Epub 2009 Mar 24. PMID 19318387
- [Background] Kosiborod M, Inzucchi SE, Krumholz HM, Masoudi FA, Goyal A, Xiao L, Jones PG, Fiske S, Spertus JA. Glucose normalization and outcomes in patients with acute myocardial infarction. Arch Intern Med. 2009 Mar 9;169(5):438-46. doi: 10.1001/archinternmed.2008.593. PMID 19273773
- [Background] Selker HP, Beshansky JR, Sheehan PR, Massaro JM, Griffith JL, D'Agostino RB, Ruthazer R, Atkins JM, Sayah AJ, Levy MK, Richards ME, Aufderheide TP, Braude DA, Pirrallo RG, Doyle DD, Frascone RJ, Kosiak DJ, Leaming JM, Van Gelder CM, Walter GP, Wayne MA, Woolard RH, Opie LH, Rackley CE, Apstein CS, Udelson JE. Out-of-hospital administration of intravenous glucose-insulin-potassium in patients with suspected acute coronary syndromes: the IMMEDIATE randomized controlled trial. JAMA. 2012 May 9;307(18):1925-33. doi: 10.1001/jama.2012.426. Epub 2012 Mar 27. PMID 22452807
- [Background] Desouza CV, Bolli GB, Fonseca V. Hypoglycemia, diabetes, and cardiovascular events. Diabetes Care. 2010 Jun;33(6):1389-94. doi: 10.2337/dc09-2082. No abstract available. PMID 20508232
- [Background] Angiolillo DJ, Fernandez-Ortiz A, Bernardo E, Ramirez C, Sabate M, Jimenez-Quevedo P, Hernandez R, Moreno R, Escaned J, Alfonso F, Banuelos C, Costa MA, Bass TA, Macaya C. Platelet function profiles in patients with type 2 diabetes and coronary artery disease on combined aspirin and clopidogrel treatment. Diabetes. 2005 Aug;54(8):2430-5. doi: 10.2337/diabetes.54.8.2430. PMID 16046311
- [Background] Alzahrani SH, Ajjan RA. Coagulation and fibrinolysis in diabetes. Diab Vasc Dis Res. 2010 Oct;7(4):260-73. doi: 10.1177/1479164110383723. Epub 2010 Sep 16. PMID 20847109
- [Background] Park KW, Park JJ, Jeon KH, Kang SH, Oh IY, Yang HM, Cho HJ, Lee HY, Kang HJ, Koo BK, Oh BH, Park YB, Kim HS. Clinical predictors of high posttreatment platelet reactivity to clopidogrel in Koreans. Cardiovasc Ther. 2012 Feb;30(1):5-11. doi: 10.1111/j.1755-5922.2010.00249.x. Epub 2010 Dec 6. PMID 21129165
- [Background] Demirtunc R, Duman D, Basar M, Bilgi M, Teomete M, Garip T. The relationship between glycemic control and platelet activity in type 2 diabetes mellitus. J Diabetes Complications. 2009 Mar-Apr;23(2):89-94. doi: 10.1016/j.jdiacomp.2008.01.006. Epub 2008 Mar 20. PMID 18358749
- [Background] Singla A, Antonino MJ, Bliden KP, Tantry US, Gurbel PA. The relation between platelet reactivity and glycemic control in diabetic patients with cardiovascular disease on maintenance aspirin and clopidogrel therapy. Am Heart J. 2009 Nov;158(5):784.e1-6. doi: 10.1016/j.ahj.2009.08.013. PMID 19853698
- [Background] Sanidas EA, Brener SJ, Maehara A, Genereux P, Witzenbichler B, El-Omar M, Fahy M, Mehran R, Gibson CM, Stone GW. Outcomes in diabetic patients undergoing primary percutaneous coronary intervention for acute anterior myocardial infarction: results from the INFUSE-AMI study. Catheter Cardiovasc Interv. 2014 Apr 1;83(5):704-10. doi: 10.1002/ccd.25203. Epub 2013 Oct 23. PMID 24030863
- [Background] Lamanna C, Monami M, Marchionni N, Mannucci E. Effect of metformin on cardiovascular events and mortality: a meta-analysis of randomized clinical trials. Diabetes Obes Metab. 2011 Mar;13(3):221-8. doi: 10.1111/j.1463-1326.2010.01349.x. PMID 21205121
- [Background] Grant PJ. Beneficial effects of metformin on haemostasis and vascular function in man. Diabetes Metab. 2003 Sep;29(4 Pt 2):6S44-52. doi: 10.1016/s1262-3636(03)72787-6. PMID 14502100
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Background] De Caterina R, Madonna R, Sourij H, Wascher T. Glycaemic control in acute coronary syndromes: prognostic value and therapeutic options. Eur Heart J. 2010 Jul;31(13):1557-64. doi: 10.1093/eurheartj/ehq162. Epub 2010 Jun 2. PMID 20519242
- [Background] Scheen AJ. DPP-4 inhibitors in the management of type 2 diabetes: a critical review of head-to-head trials. Diabetes Metab. 2012 Apr;38(2):89-101. doi: 10.1016/j.diabet.2011.11.001. Epub 2011 Dec 22. PMID 22197148
- [Background] Phung OJ, Scholle JM, Talwar M, Coleman CI. Effect of noninsulin antidiabetic drugs added to metformin therapy on glycemic control, weight gain, and hypoglycemia in type 2 diabetes. JAMA. 2010 Apr 14;303(14):1410-8. doi: 10.1001/jama.2010.405. PMID 20388897
- [Background] Karagiannis T, Paschos P, Paletas K, Matthews DR, Tsapas A. Dipeptidyl peptidase-4 inhibitors for treatment of type 2 diabetes mellitus in the clinical setting: systematic review and meta-analysis. BMJ. 2012 Mar 12;344:e1369. doi: 10.1136/bmj.e1369. PMID 22411919
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Jose T, Inzucchi SE. Cardiovascular effects of the DPP-4 inhibitors. Diab Vasc Dis Res. 2012 Apr;9(2):109-16. doi: 10.1177/1479164111436236. Epub 2012 Feb 15. PMID 22337893
- [Background] Ussher JR, Drucker DJ. Cardiovascular biology of the incretin system. Endocr Rev. 2012 Apr;33(2):187-215. doi: 10.1210/er.2011-1052. Epub 2012 Feb 8. PMID 22323472
- [Background] Scheen AJ. Cardiovascular effects of dipeptidyl peptidase-4 inhibitors: from risk factors to clinical outcomes. Postgrad Med. 2013 May;125(3):7-20. doi: 10.3810/pgm.2013.05.2659. PMID 23748503
- [Background] Rizzo MR, Barbieri M, Marfella R, Paolisso G. Reduction of oxidative stress and inflammation by blunting daily acute glucose fluctuations in patients with type 2 diabetes: role of dipeptidyl peptidase-IV inhibition. Diabetes Care. 2012 Oct;35(10):2076-82. doi: 10.2337/dc12-0199. Epub 2012 Jun 11. PMID 22688551
- [Background] Gupta AK, Verma AK, Kailashiya J, Singh SK, Kumar N. Sitagliptin: anti-platelet effect in diabetes and healthy volunteers. Platelets. 2012;23(8):565-70. doi: 10.3109/09537104.2012.721907. Epub 2012 Sep 5. PMID 22950787
- [Background] Khan S, Khan S, Imran M, Pillai KK, Akhtar M, Najmi AK. Effects of pioglitazone and vildagliptin on coagulation cascade in diabetes mellitus--targeting thrombogenesis. Expert Opin Ther Targets. 2013 Jun;17(6):627-39. doi: 10.1517/14728222.2013.764991. Epub 2013 Jan 28. PMID 23356568
- [Background] Deacon CF. Dipeptidyl peptidase-4 inhibitors in the treatment of type 2 diabetes: a comparative review. Diabetes Obes Metab. 2011 Jan;13(1):7-18. doi: 10.1111/j.1463-1326.2010.01306.x. PMID 21114598
- [Background] Barnett AH, Charbonnel B, Donovan M, Fleming D, Chen R. Effect of saxagliptin as add-on therapy in patients with poorly controlled type 2 diabetes on insulin alone or insulin combined with metformin. Curr Med Res Opin. 2012 Apr;28(4):513-23. doi: 10.1185/03007995.2012.665046. Epub 2012 Mar 1. PMID 22313154
- [Background] Frederich R, Alexander JH, Fiedorek FT, Donovan M, Berglind N, Harris S, Chen R, Wolf R, Mahaffey KW. A systematic assessment of cardiovascular outcomes in the saxagliptin drug development program for type 2 diabetes. Postgrad Med. 2010 May;122(3):16-27. doi: 10.3810/pgm.2010.05.2138. PMID 20463410
- [Background] Cobble ME, Frederich R. Saxagliptin for the treatment of type 2 diabetes mellitus: assessing cardiovascular data. Cardiovasc Diabetol. 2012 Jan 16;11:6. doi: 10.1186/1475-2840-11-6. PMID 22248301
- [Background] Monami M, Dicembrini I, Martelli D, Mannucci E. Safety of dipeptidyl peptidase-4 inhibitors: a meta-analysis of randomized clinical trials. Curr Med Res Opin. 2011 Nov;27 Suppl 3:57-64. doi: 10.1185/03007995.2011.602964. PMID 22106978
- [Background] Scirica BM, Bhatt DL, Braunwald E, Steg PG, Davidson J, Hirshberg B, Ohman P, Frederich R, Wiviott SD, Hoffman EB, Cavender MA, Udell JA, Desai NR, Mosenzon O, McGuire DK, Ray KK, Leiter LA, Raz I; SAVOR-TIMI 53 Steering Committee and Investigators. Saxagliptin and cardiovascular outcomes in patients with type 2 diabetes mellitus. N Engl J Med. 2013 Oct 3;369(14):1317-26. doi: 10.1056/NEJMoa1307684. Epub 2013 Sep 2. PMID 23992601
- [Background] Umpierrez GE, Gianchandani R, Smiley D, Jacobs S, Wesorick DH, Newton C, Farrokhi F, Peng L, Reyes D, Lathkar-Pradhan S, Pasquel F. Safety and efficacy of sitagliptin therapy for the inpatient management of general medicine and surgery patients with type 2 diabetes: a pilot, randomized, controlled study. Diabetes Care. 2013 Nov;36(11):3430-5. doi: 10.2337/dc13-0277. Epub 2013 Jul 22. PMID 23877988
- [Background] American Diabetes Association. Executive summary: Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S4-S10. doi: 10.2337/dc12-s004. No abstract available. PMID 22187471
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Scirica BM, Braunwald E, Raz I, Cavender MA, Morrow DA, Jarolim P, Udell JA, Mosenzon O, Im K, Umez-Eronini AA, Pollack PS, Hirshberg B, Frederich R, Lewis BS, McGuire DK, Davidson J, Steg PG, Bhatt DL; SAVOR-TIMI 53 Steering Committee and Investigators*. Heart failure, saxagliptin, and diabetes mellitus: observations from the SAVOR-TIMI 53 randomized trial. Circulation. 2014 Oct 28;130(18):1579-88. doi: 10.1161/CIRCULATIONAHA.114.010389. Epub 2014 Sep 4. PMID 25189213
- [Background] Engel SS, Round E, Golm GT, Kaufman KD, Goldstein BJ. Safety and tolerability of sitagliptin in type 2 diabetes: pooled analysis of 25 clinical studies. Diabetes Ther. 2013 Jun;4(1):119-45. doi: 10.1007/s13300-013-0024-0. Epub 2013 May 23. PMID 23700194
- [Background] Williams-Herman D, Round E, Swern AS, Musser B, Davies MJ, Stein PP, Kaufman KD, Amatruda JM. Safety and tolerability of sitagliptin in patients with type 2 diabetes: a pooled analysis. BMC Endocr Disord. 2008 Oct 27;8:14. doi: 10.1186/1472-6823-8-14. PMID 18954434
- [Background] Green JB, Bethel MA, Armstrong PW, Buse JB, Engel SS, Garg J, Josse R, Kaufman KD, Koglin J, Korn S, Lachin JM, McGuire DK, Pencina MJ, Standl E, Stein PP, Suryawanshi S, Van de Werf F, Peterson ED, Holman RR; TECOS Study Group. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2015 Jul 16;373(3):232-42. doi: 10.1056/NEJMoa1501352. Epub 2015 Jun 8. PMID 26052984
- [Background] McGuire DK, Van de Werf F, Armstrong PW, Standl E, Koglin J, Green JB, Bethel MA, Cornel JH, Lopes RD, Halvorsen S, Ambrosio G, Buse JB, Josse RG, Lachin JM, Pencina MJ, Garg J, Lokhnygina Y, Holman RR, Peterson ED; Trial Evaluating Cardiovascular Outcomes With Sitagliptin (TECOS) Study Group. Association Between Sitagliptin Use and Heart Failure Hospitalization and Related Outcomes in Type 2 Diabetes Mellitus: Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2016 May 1;1(2):126-35. doi: 10.1001/jamacardio.2016.0103. PMID 27437883